CLINICAL TRIAL: NCT06607887
Title: The Role of Postoperative Antibiotics in Laparoscopic Cholecystectomy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Minia University Hospital (Other)
Responsible Party: Principal Investigator, Asmaa A. Elsayed, Lecturer of clinical pharmacy, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Antibiotic77
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Infection Wound; Antibiotic Resistant Infection
Keywords: antibiotic; prophylaxis; cholecystectomy; postoperative
MeSH Terms: conditions — Wound Infection | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IV antibiotic (Experimental)
  Interventions: Drug: IV antibiotic
- Oral Antibiotic (Active Comparator)
  Interventions: Drug: Oral antibiotic

INTERVENTIONS:
Drug: IV antibiotic — Parenteral prophylactic antibiotics (cefazolin), 1st dose at the time of induction of anesthesia, 2nd dose after 12hs from the surgery.
  Arms: IV antibiotic
Drug: Oral antibiotic — Parenteral prophylactic antibiotic (cefazolin), dose at the time of induction of anesthesia and then oral antibiotic for five days postoperative.
  Arms: Oral Antibiotic

SUMMARY:
Comparison between postoperative parenteral prophylactic antibiotics, and oral antibiotics regarding the incidence of post laparoscopic cholecystectomy infection.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged above 18 years) undergoing laparoscopic cholecystectomy.

Exclusion Criteria:

* patients with comorbidities (Diabetes, malignancies, Immunosuppressed). Lost of follow-up. Patients received antibiotics within 72 hr before admission. Complicated cases involved, gangrenous and perforated cholecystitis and abscess.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-08-30 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Surgical site infection | 4 weeks
  DSSI = deep surgical site infection; SSSI = superficial surgical site infection.

SECONDARY OUTCOMES:
Fever | 4 weeks
Length of the hospital stay | 4 weeks
Hematoma and Seroma formation | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa A Elsayed, Ph.D., Principal Investigator — Sohag University
Locations (1):
- Minia University Hospital, Minya, Egypt